CLINICAL TRIAL: NCT05825443
Title: Efficacy and Safety of Postoperative Adjuvant Chemotherapy Combined With Camrelizumab for Patients With ⅡA -ⅢA Non-small Cell Lung Cancer：a Phase II , Single-arm Clinical Study
Brief Title: Adjuvant Chemotherapy Combined With Camrelizumab for ⅡA -ⅢA NSCLC Patients
Acronym: PANORAMA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2023-031
Record Dates: First submitted 2023-03-02; First posted 2023-04-24 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Immunotherapy; Chemotherapy
Keywords: Camrelizumab; Non-small Cell Lung Cancer; Adjuvant therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — camrelizumab; Cisplatin; Carboplatin; Pemetrexed

STUDY DESIGN:
Intervention Model Description: Four cycles of chemotherapy combine with camrelizumab, followed by maintenance with camrelizumab until one year or the disease progressed or unacceptable toxicity
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Patients who meet the protocol and sign the informed consent form received 4 cycles of chemotherapy combined with camrelizumab, followed by maintenance with camrelizumab until one year or the disease progressed or unacceptable toxicity. The chemotherapy regimen is decided by the researcher.
  Interventions: Drug: Camrelizumab

INTERVENTIONS:
Drug: Camrelizumab — Patients received four 21-day cycles of chemotherapy (decided by the researcher) combined with camrelizumab (200 mg in day 1), followed by maintenance with camrelizumab (200 mg in day 1, q3w), until one year or the disease progressed or unacceptable toxicity.
  Other Names: Cisplatin; carboplatin; pemetrexed; paclitaxel liposome; albumen-paclitaxel

SUMMARY:
Postoperative adjuvant chemotherapy followed by immunotherapy for non-small cell lung cancer has become a new treatment recommendation, but there are still many clinical problems to be solved in postoperative adjuvant immunotherapy. This study aims to explore the efficacy and safety of adjuvant chemotherapy combined with immunotherapy in patients with stage IIA-IIIA non-small cell lung cancer after surgery. Patients who meet the protocol and sign the informed consent form received 4 cycles of chemotherapy combined with camrelizumab, followed by maintenance with camrelizumab until one year or the disease progressed or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form before starting the study;
2. For patients with non-small cell lung cancer who have undergone surgical resection, the TNM stage after surgery is IIA-IIIA;
3. Patients cannot receive targeted adjuvant therapy;
4. 18-80 years old;
5. The patient can recover within 3-8 weeks after the operation, and receive postoperative adjuvant treatment;
6. The ECOG PS score is 0 or 1;
7. Have not received any chemotherapy for non-small cell lung cancer before enrollment;
8. Within 7 days before enrollment, the laboratory inspection must meet all the following requirements:

   * Absolute neutrophil count ≥ 1.5 × 109/L, platelet count ≥ 100 × 109/L, hemoglobin ≥ 9g/dL;
   * Total bilirubin ≤ 1.5 ULN; AST and ALT ≤ 2.5 ULN;
   * Serum creatinine ≤ 1.25 ULN, or serum creatinine clearance ≥ 60ml/min;
9. Female patients must meet: menopause or have undergone surgical sterilization. Women with fertility must take effective contraceptive measures. Do not breastfeed.
10. Male patients must agree to use appropriate contraceptive measures.

Exclusion Criteria:

1. Known or suspected to be allergic to the drug or any component of the drug related to the test;
2. Patients who can receive targeted treatment;
3. Other malignant tumors in five years before enrollment, excluding the cured cervical carcinoma in situ, the cured skin basal cell carcinoma, and other types of tumors that were cured only after surgical treatment;
4. Myocardial infarction, unstable angina pectoris and grade II congestive heart failure in six months before enrollment; New angina pectoris occurred within 3 months; Ventricular arrhythmia requiring medication;
5. Uncontrolled hypertension after treatment with antihypertensive drugs, i.e. systolic blood pressure ≥ 140mmHg or diastolic blood pressure ≥ 90mmHg;
6. History of HIV infection, active period of HCV infection, active period of HBV infection (HBV-DNA>1000 copies/ml);
7. The researcher judged that there was a risk of bleeding;
8. Active severe clinical infection (≥ grade 3 CTCAE V5.0);
9. Epilepsy patients who need medication;
10. Allogeneic organ transplantation;
11. Patients who need kidney dialysis;
12. Thrombotic or embolic venous or arterial events occurred within six months before enrollment;
13. Serious uncured wounds, ulcers or fractures;
14. Interstitial pneumonia;
15. Any malabsorption disease;
16. Any disease that is unstable or may endanger the patient's safety;
17. Drug abuse, medical, psychological or social diseases;
18. Participate in other clinical studies within 3 months before enrollment;
19. During pregnancy or lactation;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Two-years disease free survival (2y-DFS) | Up to approximately 2 years
  DFS, defined as the time from first dose of Camrelizumab to the first occurrence of disease recurrence as determined by the investigator with use of RECIST v1.1 or death from any cause, whichever occurs first. According to the K-M curve, the proportion of disease-free progression in 2 years.

SECONDARY OUTCOMES:
Three-years disease free survival (3y-DFS) | Up to approximately 3 years
  According to the K-M curve, the proportion of disease-free progression in 3 years
Five-years disease free survival (5y-DFS) | Up to approximately 5 years
  According to the K-M curve, the proportion of disease-free progression in 5 years
Disease free survival (DFS） | Up to approximately 2 years
  DFS, defined as the time from first dose of Camrelizumab to the first occurrence of disease recurrence as determined by the investigator with use of RECIST v1.1 or death from any cause, whichever occurs first.
Overall survival (OS) | Up to approximately 5 years
  Defined as the time from randomization to death from any cause.
Two-years overall survival（2y-OS) | Up to approximately 2 years
  According to the K-M curve, the proportion of OS in 2 years
Three-years overall survival（3y-OS) | Up to approximately 3 years
  According to the K-M curve, the proportion of OS in 3 years
Five-years overall survival（5y-OS) | Up to approximately 5 years
  According to the K-M curve, the proportion of OS in 5 years
Treatment-related adverse events（TRAE） | Up to approximately 1 year
  The incidence of TRAE and the incidence of level 3-4 TRAE according to CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guandong, Guangdong, China

IPD SHARING:
Plan to Share IPD: No